CLINICAL TRIAL: NCT01073670
Title: Quantification of Postoperative Coagulation Following Administration of Indomethacin to Expedite Fast-tracking of Cardiac Surgical Patients
Brief Title: Indomethacin and Cardiac Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Dr. Joel Parlow, Head, Department of Anesthesiology & Perioperative Medicine, Queen's University and Kingston General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ANAE-062-00
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Hemorrhage
Keywords: NSAIDs; bleeding; thromboelastography; cardiac surgery; Indomethacin; acetaminophen
MeSH Terms: conditions — Hemorrhage | interventions — Indomethacin; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acetaminophen (Active Comparator): Participants received a loading dose of acetaminophen (2600 mg) at induction followed by 1300 mg at 6, 12, 18 and 24 hours following cardiac bypass surgery.
  Interventions: Drug: Acetaminophen
- Indomethacin (Experimental): Participants were given 100 mg of indomethacin at induction and then 50 mg at 6, 12, 18 and 24 hours following cardiac bypass surgery.
  Interventions: Drug: Indomethacin
- Combination (Experimental): Participants were given a loading dose of 1300 mg of acetaminophen and 50 mg of Indomethacin followed by 650mg of acetaminophen and 25 mg of indomethacin at 6, 12, 18 and 24 hours following cardiac bypass surgery.
  Interventions: Drug: Acetaminophen & Indomethacin

INTERVENTIONS:
Drug: Indomethacin — Indomethacin was given via suppository at time of induction for anesthesia (2 x 50 mg) followed by one 50 mg suppository at 6, 12, 18 and 24 hours following cardiac bypass surgery.
  Other Names: Indocin
  Arms: Indomethacin
Drug: Acetaminophen & Indomethacin — Subjects were given a loading dose of acetaminophen (1300 mg) and indomethacin (50 mg)by suppository at the time of induction for anesthesia and then given 650mg acetaminophen + 25 mg indomethacin at 6, 12, 18 and 24 hours following cardiac bypass surgery.
  Other Names: Tylenol; Indocin
  Arms: Combination
Drug: Acetaminophen — Subjects were given a loading dose of 2600 mg of acetaminophen (via suppository) at time of induction for anesthesia then given 1300mg at 6, 12, 18 and 24 hours following cardiac bypass surgery.
  Other Names: Tylenol
  Arms: Acetaminophen

SUMMARY:
Following signed informed consent, patients scheduled for elective cardiac surgery were randomly assigned to one of 3 groups to be given acetaminophen, Indomethacin or a combination of both immediately following induction and then at 6, 12, 18 & 24 hours following surgery. Our primary outcome measure was the amount of blood drained from the mediastinal tubes and chest drains. Secondary outcome measures included conventional blood coagulation indices as well as other measures of clotting as indicated by thromboelastography (TEG). Other secondary outcome measures included consumption of morphine equivalents and pain scores.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo either elective coronary artery bypass or single valve replacement
* normal platelet count
* normal prothrombin time
* normal partial thromboplastin time
* normal serum creatinine

Exclusion Criteria:

* sensitivity to study drugs
* history of bleeding diathesis
* renal dysfunction
* active peptic ulcer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2000-08; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
amount of blood lost via chest drains during and following cardiac bypass surgery | during surgery and then until chest drains removed (< 24 hours)

SECONDARY OUTCOMES:
blood clotting indices (i.e., conventional and using thromboelastography) | perioperative period until 24 hours post-operative
Morphine equivalents required to provide effective analgesia | perioperative period until 24 hours post-operative
  The milligram quantities of morphine or the equivalents of morphine administered (in addition to the acetaminophen, indomethacin or combination therapy) were recorded and compared between groups. This provided an indication of how effective each of our interventions were at providing pain relief.
pain scores | perioperative period until 24 hours post-operative
  Resting pain scores were recorded for all subjects at 6, 12 18 and 24 hours following surgery and compared between groups. These scores provided an indication as to the efficacy of each of our interventions at providing pain relief.

CONTACTS AND LOCATIONS:
Overall Officials: Joel L Parlow, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada